CLINICAL TRIAL: NCT03794596
Title: A Proof of Concept, Window Trial of the IMmunological Effects of AveLumab and Aspirin in Triple-Negative Breast Cancer
Acronym: IMpALA
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: IP breach
Sponsor: The Christie NHS Foundation Trust (Other)
Collaborators: University of Manchester (Other)
Responsible Party: Principal Investigator, Rachel Cox, Non CI _Project manager, The Christie NHS Foundation Trust
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CFT/sp123; 2018-004121-80 (EudraCT Number); 16_DOG02_289 (Other: Sponsor Local Identifier); 017NovCC1079 (Other Grant/Funding Number: Breast Cancer Now)
Record Dates: First submitted 2018-11-22; First posted 2019-01-07 (Actual); Last update posted 2019-07-22 (Actual); Status verified 2019-07

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — avelumab; Aspirin; Lansoprazole; Proton Pump Inhibitors

STUDY DESIGN:
Intervention Model Description: Patients will be randomly assigned to one of two arms:-
  * 21 patients into Arm A: Avelumab + Proton Pump Inhibitor (PPI)
  * 21 patients into Arm B: Avelumab + Aspirin + PPI
Who Masked: Outcomes Assessor
Masking Description: Laboratory staff and the blinded statistician will remain blinded to trial treatment arm
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- (Arm A) Avelumab + PPI (Experimental): 21 patients into Arm A: Avelumab + Proton Pump Inhibitor (PPI)
  Interventions: Drug: Avelumab; Drug: Lansoprazole (Proton Pump Inhibitor)
- (Arm B) Avelumab + Aspirin + PPI (Experimental): 21 patients into Arm B: Avelumab + Aspirin + PPI
  Interventions: Drug: Avelumab; Drug: Aspirin; Drug: Lansoprazole (Proton Pump Inhibitor)

INTERVENTIONS:
Drug: Avelumab — Colourless odourless aqueous solution for infusion at dose of 10mg/kg
  Other Names: Bavencio
Drug: Aspirin — 300mg tablets
  Arms: (Arm B) Avelumab + Aspirin + PPI
Drug: Lansoprazole (Proton Pump Inhibitor) — 300mg capsule
  Other Names: Lansoprazole

SUMMARY:
This research is being done because the investigators are looking for new and better ways to treat a type of breast cancer called triple negative breast cancer. This type of breast cancer can be more difficult to treat than other types of breast cancer as it does not respond to drugs such as hormonal therapies. One type of treatment that looks promising is immunotherapy using new drugs called immune checkpoint inhibitors.

Immune checkpoints help to regulate the immune system and can stop the immune system from attacking cancer cells. Immune checkpoint inhibitors block this 'off-switch' and aim to help the immune system control the cancer. These drugs have been very effective in other cancers such as melanoma and are now being tested in breast cancer.

In this study patients will receive an immune checkpoint inhibitor called avelumab. Half the patients on the study will also receive aspirin tablets for approximately 18 days as the investigators wish to compare the effects of avelumab alone versus in combination with aspirin.

Patients will attend hospital approximately five times in order to complete all necessary study assessments. The first visit screens patients for suitability, after which a baseline visit will collect the first of two breast tissue biopsies. At the third visit a single dose of Avelumab will be given via an infusion (a drip in the forearm). Patients will then return approximately two weeks later for a second breast tissue biopsy before having a final follow up visit another two weeks later. Blood and urine samples will be taken at various visits throughout the study to help us learn more about the effects these treatments may have on the immune system and on breast cancer cells.

DETAILED DESCRIPTION:
TNBC is an aggressive subtype of breast cancer associated with poor survival and new treatments are needed. A key feature of cancer is its ability to go undetected by the immune system. Recent developments in cancer research have identified immune checkpoints as a possible treatment option as they seem to promote an anti-tumour immune response.

Some breast cancers have considerable cancer cell infiltration, which has been associated with better prognosis. This is where white blood cells have permeated the cancer cell and infiltrated the infected cell in an attempt to 'cure' the infected cell. Greater immune-sensitivity is thought to correlate with greater cancer cell infiltration therefore researchers are looking at ways in which immune-sensitivity can be improved.

One approach is to target inflammation that is known to play a major role in cancer development and progression. Certain proteins can often be abnormally expressed in many cancers. In preclinical models the investigators recently demonstrated that the presence of certain cancer cell-derived proteins is critical for the growth of tumours formed by melanoma, colorectal and breast mouse cancer cell lines. In the mouse preclinical trials it indicated that by blocking the cancer cells ability to produce these proteins was associated with a marked shift in the inflammatory profile. To test this theory, this study will use aspirin as the chosen protein inhibitor and it is speculated that the addition of aspirin might enhance the efficacy of the immune checkpoint blockade, avelumab.

TRIAL AIMS & DESIGN

The aim of this trial is to determine whether aspirin enhances the efficacy of avelumab by promoting a greater anti-cancer immune response. This is a multi-centre study recruiting patients with confirmed TNBC from across four trial sites within the United Kingdom. It is anticipate that 50 participants will need to be screened in order to successfully enrol 42 patients onto the trial. Patients will be randomly assigned to one of two arms:-

* 21 patients into Arm A: Avelumab + Proton Pump Inhibitor (PPI)
* 21 patients into Arm B: Avelumab + Aspirin + PPI

The estimated duration of participation for a participant is up to 10 weeks. Each subject will be asked to complete 5 study visits. After successfully completing a Screening Visit (Visit 1), each eligible subject will attend for a Baseline Visit (Visit 2) and will be randomly assigned to treatment ARM A or ARM B. As part of the baseline visit subjects will have their first of two breast tumour biopsies. All subjects will commence their PPI following the baseline visit, those subjects randomised to ARM B will also commence their Aspirin at this time. At visit 3 all subjects will receive their Avelumab infusion. At Visit 4 (Follow up Visit A) each subject will undergo their second research biopsy and further research blood sampling this will be the first of two follow up visits, with Visit 5 (Follow up Visit B) concluding the patients participation.

Visit windows have been used to aid visit planning in the hope that most research appointments can take place in line with patients' ordinary care visits so as to reduce any burden inflicted on the patient.

Adverse events (AEs) and Serious Adverse Events (SAEs) will be collected from the time of randomisation and will continue to be collected up until Visit 5 (Follow up Visit B). All post biopsy treatment will be at the discretion of the subject's treating physician per local standard of care.

PATIENT IDENTIFICATION & SCREENING

The study will be conducted as a multi-centre trial consisting of four NHS secondary care out-paints clinics from across the United Kingdom. Each site has been chosen for their expertise in oncology and their ability to identify patients for the trial directly from their clinics with each centre treating between 20 to 40 patients per annum; this pool of patients will constitute the source of recruitment in the study, PIC sites may also be used.

Potential participants will be identified by the Principal Investigators multi-disciplinary team following recent diagnosis of TNBC. The multidisciplinary team shall be trained on the study protocol and required to sign the trial delegation and training log in advance of working on the trial or identifying participants. Potential participants will have at least 24 hours to read the patient information and decide if they would like to participate in the study. Participants must have the capacity to provide fully informed consent. Participants must not participate in any other therapeutic trials whilst on study treatments, however once all study treatments as specified by trial schema are completed, participation in further studies will not be affected.

At the screening visits the following data will be collected:-

* Informed consent
* Demographics
* Medical history
* Concomitant medication
* Complete Physical examination
* Vital Signs
* 12-lead Electrocardiograph (ECG)
* ECOG performance status
* Blood tests:-

  * Biochemistry: AST or ALT, LDH, Alk Phos, total bilirubin, sodium, potassium, urea, creatinine, total protein, albumin, adjusted calcium
  * Haematology: FBC: Hb, Platelets, ANC, WBC, Lymphocytes, basophils, eosinophils
  * Thyroid Function: Free T4, TSH
  * Urinalysis
* Pregnancy testing
* Optional: Microbiome samples kit dispensation (Stool sample, Saliva sample, Nasal Swab)
* Baseline tumour assessment

BASELINE VISIT

The following assessments will be conducted at the time of this visit:

* Adverse Events
* Concomitant medication
* Vital Signs
* ECOG performance status
* Eligibility
* Randomisation
* Research Bloods (Circulating tumour DNA (CtDNA); Plasma for Cytokine Analysis; PBMC extraction for immunophenotyping)
* Mid-stream Urine sample for prostaglandin
* Optional: Microbiome samples kit collection (Stool sample, Saliva sample, Nasal Swab)
* Breast Tissue Biopsy
* Pre-treatment dispensation (Arm A: PPI OR Arm B: PPI + aspirin)
* Diary card training and dispensation
* Pre-treatment Reminder Telephone call
* TREATMENT & FOLLOW UP VISITS

Visit 3: I.V visit

The following assessments will be conducted at the time of this visit:

* Assessment of Adverse Events
* Concomitant medication
* Vital Signs
* *Laboratory tests *(Biochemistry, Haematology and Urinalysis only if screening labs were >14 day prior to visit 3)
* **Pregnancy testing **(only if screen pregnancy test was >14days prior to day Visit 3)
* Microbiome samples kit dispensation only (Stool, Saliva, Nasal Swab )
* Mid-stream Urine sample for prostaglandin
* Diary card - Pre-treatment compliance check (Arm A: PPI, Arm B: PPI + aspirin)
* Avelumab (10mg/kg i.v.)

Visit 4: Follow up A The following assessments will be conducted at the time of this visit

* Adverse Events
* Concomitant medication
* Research Bloods (CtDNA); Plasma for Cytokine Analysis; Immunophenotyping)
* Microbiome sample kit collection (Stool sample, Saliva sample, Nasal Swab)
* Mid-stream Urine sample for prostaglandin
* Breast Tumour Biopsy
* Diary card - Pre-treatment compliance check (Arm A: PPI, Arm B: PPI + aspirin)

Visit 5: Follow up B

The following assessments will be conducted at the time of this visit:

* Adverse Events
* Concomitant medication
* Symptom Directed Physical examination
* Vital Signs (BP, HR, Sp02, Temp)
* ECOG performance status
* Laboratory blood tests

  * Biochemistry: AST or ALT, LDH, Alk Phos, total bilirubin, sodium, potassium, urea, creatinine, total protein, albumin, adjusted calcium
  * Haematology: FBC - Hb, Platelets, ANC, WBC, Lymphocytes, basophils, eosinophils
  * Thyroid Function: Free T4, TSH
  * Urinalysis
* Research Bloods (CtDNA); Plasma for Cytokine Analysis; Immunophenotyping)

SAFETY REVIEW An Independent Trial Steering Committee (TSC) and Data Monitoring Committee (IDMC) is being formed and will review trial safety data as a combined committee group.

TRANSLATIONAL RESEARCH With consent the following samples will be collected from patients and held by the Manchester Cancer Research

Centre (MCRC) biobank:

* Microbiome samples
* Research blood samples
* Breast Tissue Biopsies

The MCRC biobank holds a generic research tissue bank ethics approval under their HTA license and will release the samples for relevant research, subject to approval by the Biobank's Access Committee.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent, willing and able to comply with the trial protocol for the duration of the trial including all treatments and scheduled biopsies.
2. Female patients, age 18 and over
3. Histologically confirmed triple negative invasive breast cancer as defined as oestrogen receptor (ER) negative, progesterone receptor (PgR) negative (if available, otherwise PgR unknown), (as defined by Allred score 0- 2 or <1% of tumour cells positive for stain) and HER2 negative (immunohistochemistry 0/1+ or negative by in situ hybridization) as determined by local laboratory. Have previously untreated, non-metastatic TNBC with a tumour amenable to multiple biopsies including a T stage of at least T2. Note multifocal primary tumours are allowed providing at least one tumour meets the criteria above. All biopsies should be obtained from the same tumour.
4. Have previously untreated, non-metastatic TNBC with a tumour amenable to multiple biopsies including a T stage of at least T2. Note multifocal primary tumours are allowed providing at least one tumour meets the criteria above. All biopsies should be obtained from the same tumour.
5. ECOG performance status 0/1
6. Women of childbearing potential (WOCBP), defined as not surgically sterilized or not post-menopausal for at least 24 months if age ≤55 years or 12 months if age >55 years, must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 14 days prior to the start of either IMP study treatment (Avelumab, and Aspirin if applicable).
7. Adequate organ function:-

   1. Adequate Hepatic function:

      * AST and ALT <2.5x ULN
      * Alkaline phosphatase ≤2 x ULN
      * Total Bilirubin within normal range i.e. ≤1.5 x ULN. If AST/ALT and Alkaline phosphatase are within normal limits then isolated elevation of bilirubin to 3≤ ULN and a presumptive diagnosis of Gilbert's syndrome is permitted.
   2. Adequate organ function as defined by:

      * Bone marrow function: Hb ≥100g/L
      * Absolute neutrophil count ≥1.5 x 109/L
      * Platelets ≥100 x 109/L
      * Hemoglobin >9 g/dL
      * Renal function: Creatinine ≤1.5 x ULN OR > 50ml/min using the Cockcroft-Gault formula (appendix 4).

Exclusion Criteria:

Patients meeting any of the following criteria must not be enrolled in the study:

1. Prior systemic anti-cancer treatment (immune therapy, targeted therapy, vaccine therapy, or investigational treatment) for triple negative breast cancer.
2. Current use of a prohibited medication as described in section 7.11.
3. Malignancy within the last 5 years except: adequately treated non-melanoma skin cancer; curatively treated in situ cancer of the cervix, ductal carcinoma in situ (DCIS); stage 1, grade I endometrial carcinoma.
4. Has received a live vaccine within 30 days of the first dose of study treatment.

   NB Seasonal influenza vaccines are generally inactivated flu vaccines and are allowed; intranasal influenza vaccines (eg FluMist®) are live attenuated vaccines and are not allowed.
5. Contraindications to aspirin dosing including hypersensitivity to aspirin (eg known aspirin sensitive asthma; history of peptic ulcer disease, gastric bleeding or cerebrovascular haemorrhages; haemorrhagic diathesis.
6. Evidence of distant metastases apparent prior to randomisation. Patients who are diagnosed with distant metastases during the course of the study can complete study procedures if willing to do so.
7. Significant cardiovascular disease including a history of myocardial infarction, acute coronary syndrome or coronary angioplasty/stenting/bypass grafting within the last 6 months or clinically significant congestive heart failure.
8. Any other serious or unstable pre-existing medical conditions (aside from malignancy exceptions specified above), psychiatric disorders, or other conditions that in the opinion of the investigator could interfere with the patient's safety, obtaining informed consent, or compliance with study procedures.
9. Known Human Immunodeficiency Virus (HIV), Hepatitis B Virus (HBV), or Hepatitis C Virus (HCV) infection (patients with laboratory evidence of cleared or chronic (not active) HBV and HCV infection will be permitted).
10. Patients with active, known or suspected autoimmune disease. Patients with type 1 diabetes mellitus, hypothyroidism only requiring hormone replacement, skin or rheumatological disorders (such as vitiligo, psoriasis, rheumatoid arthritis or alopecia) not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger will be permitted to enrol. Autoimmune conditions such as ulcerative colitis that have been definitively treated (e.g. with total colectomy) will be permitted to enrol but should be discussed with the CI.
11. Patients with a condition requiring systemic treatment with either corticosteroids (>10 mg daily prednisone equivalent) or other immunosuppressive medications within 14 days of study drug administration. Inhaled or topical steroids and adrenal replacement steroid doses > 10 mg daily prednisone equivalent are permitted in the absence of active autoimmune disease.
12. Patients with interstitial lung disease that is symptomatic or may interfere with the detection or management of suspected drug-related pulmonary toxicity.
13. Patients unable to swallow orally administered medication and patients with gastrointestinal disorders likely in to interfere with absorption of the trial medication.
14. Females who are pregnant or breast-feeding.
15. Active infection requiring systemic treatment.
16. Current or previous regular use of aspirin (at any dose) or current use of another NSAID for any indication (see appendix IV for list of medications not permitted in the trial). Regular aspirin use is defined as taking aspirin more than twice in any given week for more than 4 consecutive weeks. Current NSAID use is defined as taking any NSAID for more than a week in the preceding month. If investigators feel that this definition may unfairly exclude a participant, this can be discussed with the CI/MCTU and a case by case decision will be made.
17. Known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to the study treatments.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female patients, age 18 and over
Enrollment: 0 (Actual)
Dates: Start 2019-09 (Estimated); Primary Completion 2021-02-28 (Estimated); Study Completion 2021-02-28 (Estimated)

PRIMARY OUTCOMES:
Mean combined gene expression of COX-2 tumour-promoting genes | 7 weeks
  Mean combined gene expression of COX-2 tumour-promoting genes, in samples taken post treatment

SECONDARY OUTCOMES:
Post treatment tumour infiltrating lymphocytes (TIL) | 7 weeks
  Post treatment tumour infiltrating lymphocytes (TIL) assessed by IHC using standardised methodology (Salgado et al., 2015)
Mean combined gene expression of the elements of the denominator of the COX-2 ratio | 7 weeks
  Mean combined gene expression of the elements of the denominator of the COX-2 ratio, in samples taken post treatment.
The post treatment COX-2 ratio | 7 weeks
  The post treatment COX-2 ratio (a ratio of mean expression of 9 tumour-promoting to 15 tumour-inhibitory genes)
Safety and tolerability assessed by grade 3-4 AEs and SAEs | 7 weeks
  Safety and tolerability assessed by grade 3-4 AEs and SAEs. In addition, grade 2 renal toxicity AEs (creatinine rise) and grade 2 gastrointestinal toxicity AEs (duodenal perforation, dyspepsia, oesophageal haemorrhage, dysphagia, oesophageal pain, oesophageal perforation, oesophagitis).

CONTACTS AND LOCATIONS:
Overall Officials: Anne Armstrong, Principal Investigator — The Christie NHS Foundation Trust

IPD SHARING:
Plan to Share IPD: No